CLINICAL TRIAL: NCT04025138
Title: Fatigability Compared Men and Women Induced According to the Distance Traveled on an Ultra-marathon in the Mountains
Acronym: UTMB_2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19CH060; 2019-A00736-51 (Other: ANSM)
Record Dates: First submitted 2019-07-03; First posted 2019-07-18 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Ultra-marathon Runners
Keywords: Sex differences; Ultra-endurance running; Mont Blanc Ultra Trail; Transcranial Magnetic Stimulation (TMS); Neuromuscular tests; Plantar flexors; Knee extensors; Force/Velocity Profile (FVP)
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- female subjects involved in races over 100 km (F>100) (Experimental): Female subjects involved in races over 100 km (F>100) will be included. They will have neuromuscular tests in isometric mode, Transcranial Magnetic Stimulation (TMS), neuromuscular fatigue assessment test, treadmill, blood sample and urinary sample.
  Interventions: Other: Neuromuscular tests in isometric mode; Device: Transcranial Magnetic Stimulation (TMS); Other: Neuromuscular fatigue assessment test; Other: treadmill; Biological: Blood sample; Biological: Urinary sample
- female subjects involved in races less than 60 km (F<60) (Experimental): Female subjects involved in races less than 60 km (F<60) will be included. They will have neuromuscular tests in isometric mode, Transcranial Magnetic Stimulation (TMS), neuromuscular fatigue assessment test, treadmill, blood sample and urinary sample.
  Interventions: Other: Neuromuscular tests in isometric mode; Device: Transcranial Magnetic Stimulation (TMS); Other: Neuromuscular fatigue assessment test; Other: treadmill; Biological: Blood sample; Biological: Urinary sample
- male subjects involved in races over 100 km (H>100) (Experimental): Male subjects involved in races over 100 km (H>100) will be included. They will have neuromuscular tests in isometric mode, Transcranial Magnetic Stimulation (TMS), neuromuscular fatigue assessment test, treadmill, blood sample and urinary sample.
  Interventions: Other: Neuromuscular tests in isometric mode; Device: Transcranial Magnetic Stimulation (TMS); Other: Neuromuscular fatigue assessment test; Other: treadmill; Biological: Blood sample; Biological: Urinary sample
- male subjects involved in races less than 60 km (H<60) (Experimental): Male subjects involved in races less than 60 km (H<60) will be included. They will have neuromuscular tests in isometric mode, Transcranial Magnetic Stimulation (TMS), neuromuscular fatigue assessment test, treadmill, blood sample and urinary sample.
  Interventions: Other: Neuromuscular tests in isometric mode; Device: Transcranial Magnetic Stimulation (TMS); Other: Neuromuscular fatigue assessment test; Other: treadmill; Biological: Blood sample; Biological: Urinary sample

INTERVENTIONS:
Other: Neuromuscular tests in isometric mode — Protocol for neuromuscular tests in isometric mode will be assessed by the composite of these measures :
  * Voluntary maximum forces plantar flexors and knee extensors
  * Electrically evoked forces
  * ElectroMyoGraphic activity (EMG)
  * Three-Modality Evoked Potentials (TMEPs)
Device: Transcranial Magnetic Stimulation (TMS) — Measure of supraspinal activation level and cortical excitation by Transcranial Magnetic Stimulation (TMS).
Other: Neuromuscular fatigue assessment test — Neuromuscular fatigue assessment test in dynamic mode will be assessed by the Force/Velocity Profile (FVP) measure: 2 sprints of 8 seconds on a cycle ergometer.
Other: treadmill — 2 sessions of treadmill will be realized: 8 and 10 km.h-1 for level running and 7 km.h-1 with 10% slope for graded running.
Biological: Blood sample — Blood sample will be realized to measure hemorrheologic and hematologic parameters.
Biological: Urinary sample — Urinary sample will be realized to measure hemorrheologic and hematologic parameters.

SUMMARY:
Acute physiological consequences of ultra-marathon running are still unknown, particularly in women. Some studies have suggested that the proportion of fatigue attributable to peripheral and central mechanisms varies between males and females; however, results are contradictory.

The results from the investigators of the present experiment in two studies conducted in 2009 and 2012 showed that:

* A large part of fatigue induced by a mountain ultra-marathon could be attributed to central fatigue in males and that,
* Females exhibited less peripheral fatigue in the plantar flexors than males did after a 110-km ultra-trail-running race.

According to the literature, there seems to be a plateau in fatigue after 12-15 hours of running.

DETAILED DESCRIPTION:
Thus, the main purpose of the present project is to investigate whether sex differences in neuromuscular fatigue in plantar flexors depend on the distance (> 100 km vs < 60 km).

ELIGIBILITY:
Inclusion Criteria:

* Subject listed in the race "2019 Mont Blanc Ultra Trail"
* Affiliates or beneficiaries of social security scheme
* Signed consent

Exclusion Criteria:

* Subject having been injured in the previous 3 months
* Pregnant woman
* Chronic joint diseases
* Chronic or central neurological pathologies
* Taking neuroactive substances that can alter corticospinal excitability
* Contraindication to experimental procedures including Transcranial Magnetic Stimulation (TMS)
* Taking corticosteroids in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Variation (%) of the amplitudes of the electric shock | 5 or 6 day before the race and 1 hour after
  Measured by the electrically evoked force after contraction in isometric mode of the plantar flexors

SECONDARY OUTCOMES:
Voluntary maximum forces plantar flexors | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Measured by voluntary maximum forces plantar flexors test (seat type Cybex) in percentage (%).
Voluntary maximum forces knee extensors | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Voluntary maximum forces knee extensors measures by seat type Cybex in percentage (%).
Electrically evoked forces | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Electrically evoked forces measures by neurostimulator in percentage (%).
ElectroMyoGraphic activity (EMG) | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  ElectroMyoGraphic activity (EMG) measures by electromyography. The EMG signal will be recorded with pairs of electrodes fixed with an adhesive tape bilaterally over the muscular belly.
Three-Modality Evoked Potentials (TMEPs) | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Three-Modality Evoked Potentials (TMEPs) measures by magnetic stimulator in percentage (%).
Transcranial Magnetic Stimulation (TMS) | 5 or 6 day before the race and 1 hour after
  Analysis :
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Measured supraspinal activation level and cortical excitation by Transcranial Magnetic Stimulation (TMS) in percentage (%).
Force/Velocity Profile (FVP) | 5 or 6 day before the race and 1 hour after
  Analysis:
  * Quantification of neuromuscular fatigue assessment;
  * Evolution of race mechanics and the energy cost between males and females depending on the distance of the race.
  Measured Force/Velocity Profile (FVP) test: 2 sprints of 8 seconds on a cycle ergometer.
Blood viscosity | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
Number of red blood cell | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
Number of platelets | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
Number of white blood cells | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
Rate of hemoglobin (%) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
creatinine (mg/L) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
C reactive protein (CRP) (mg/L) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
urea (g/L) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
uric acid (mg/L) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
lactate (mg/L) | 5 or 6 day before the race and 1 hour after
  Measured by blood sample.
Proteinuria-density urinary (mg/24h) | 5 or 6 day before the race and 1 hour after
  Measured by urinary sample.
Kinematic variable | 5 or 6 day before the race and 1 hour after
  Measured by treadmill result.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Guillaume MILLET, PhD, Study Director — University of Saint-Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robert M, Stauffer E, Nader E, Skinner S, Boisson C, Cibiel A, Feasson L, Renoux C, Robach P, Joly P, Millet GY, Connes P. Impact of Trail Running Races on Blood Viscosity and Its Determinants: Effects of Distance. Int J Mol Sci. 2020 Nov 12;21(22):8531. doi: 10.3390/ijms21228531. PMID 33198320
- [Result] Temesi J, Besson T, Parent A, Singh B, Martin V, Brownstein CG, Espeit L, Royer N, Rimaud D, Lapole T, Feasson L, Millet GY. Effect of race distance on performance fatigability in male trail and ultra-trail runners. Scand J Med Sci Sports. 2021 Sep;31(9):1809-1821. doi: 10.1111/sms.14004. Epub 2021 Jul 12. PMID 34170574
- [Result] Foure A, Besson T, Stauffer E, Skinner SC, Bouvier J, Feasson L, Connes P, Hautier CA, Millet GY. Sex-related differences and effects of short and long trail running races on resting muscle-tendon mechanical properties. Scand J Med Sci Sports. 2022 Oct;32(10):1477-1492. doi: 10.1111/sms.14203. Epub 2022 Jul 6. PMID 35730335
- [Result] Pastor FS, Besson T, Varesco G, Parent A, Fanget M, Koral J, Foschia C, Rupp T, Rimaud D, Feasson L, Millet GY. Performance Determinants in Trail-Running Races of Different Distances. Int J Sports Physiol Perform. 2022 Jun 1;17(6):844-851. doi: 10.1123/ijspp.2021-0362. Epub 2022 Feb 25. PMID 35213820
- [Result] Sabater Pastor F, Varesco G, Besson T, Koral J, Feasson L, Millet GY. Degradation of energy cost with fatigue induced by trail running: effect of distance. Eur J Appl Physiol. 2021 Jun;121(6):1665-1675. doi: 10.1007/s00421-021-04624-5. Epub 2021 Mar 5. PMID 33666727
- [Derived] Trama R, Blache Y, Hintzy F, Rossi J, Millet GY, Hautier C. Does neuromuscular fatigue generated by trail running modify foot-ground impact and soft tissue vibrations? Eur J Sport Sci. 2023 Jul;23(7):1155-1163. doi: 10.1080/17461391.2022.2093649. Epub 2022 Jul 10. PMID 35730761
- [Derived] Besson T, Parent A, Brownstein CG, Espeit L, Lapole T, Martin V, Royer N, Rimaud D, Sabater Pastor F, Singh B, Varesco G, Rossi J, Temesi J, Millet GY. Sex Differences in Neuromuscular Fatigue and Changes in Cost of Running after Mountain Trail Races of Various Distances. Med Sci Sports Exerc. 2021 Nov 1;53(11):2374-2387. doi: 10.1249/MSS.0000000000002719. PMID 34107510